CLINICAL TRIAL: NCT01139541
Title: Testing Strategies for Increasing Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Collaborators: Blue Cross Blue Shield (Other)
Responsible Party: Principal Investigator, Michael Norton, Associate Professor, Harvard University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: WalkStation1
Record Dates: First submitted 2010-06-03; First posted 2010-06-08 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Sedentary Lifestyle; Obesity
MeSH Terms: conditions — Sedentary Behavior; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention): Participants in the control condition will be asked to refrain from using the WalkStations during the study period.
- Individual (Experimental): In the individual condition, participants will not be part of a team. They will receive weekly email feedback on their Walkstation performance (e.g. number of time slots they signed up for, and number of times they showed up for the time slot.)
  Interventions: Behavioral: Social walking intervention
- Pairs (Experimental): In the pair condition, participants will be randomly assigned to a partner. They will receive the same feedback as those in the individual condition, for both themselves AND their partner.
  Interventions: Behavioral: Social walking intervention
- Groups (Experimental): In the group condition, participants will be randomly assigned to a group of 5 people. They will receive the same feedback as those in the individual condition, for both themselves AND each member of their group.
  Interventions: Behavioral: Social walking intervention

INTERVENTIONS:
Behavioral: Social walking intervention — In this intervention, we are interested in the impact of group dynamics on the propensity to use the Walkstations. The intervention consists of 4 levels: control, individual, pair, and group.
  Arms: Groups; Individual; Pairs

SUMMARY:
The purpose of the study is to learn more about effective ways to motivate people to increase their non-exercise energy expenditure exercise. This is an important research question because obesity and weight-related issues are increasingly becoming a problem in America. This project will address this research question by testing the effect of group dynamics in motivating employees who are predominantly sedentary to use Walkstations at work. The Walkstations are treadmills that move at a very slow rate (maximum 2miles / hour) and are attached to a work station (i.e. with computer and telephone); they therefore are designed to increase energy spent not through heavy exercise, but through small changes in posture and movement associated with routines in daily life (called nonexercise activity thermogenesis or NEAT). The proposed study is designed to build upon previous research (Levine et al., 2005) suggesting the role of NEAT-enhanced behaviors in weight loss.

In this study, the investigators are interested in the impact of group dynamics on the propensity to use the Walkstations. Participants in the active arms will be asked to use the Walkstations for at least 3 hours per week. They will do so by signing up for a time slot. During their session, they will be asked to log into the scheduling system to indicate that they are using the Walkstation. Walkstation usage will be assessed by log-in data: employees will log-in to the phone and computer when they use the Walkstation. This log-in data is work-station specific; therefore the investigators will be able to tell when a given subject used the Walkstation.

Subjects will be randomly assigned to one of three conditions:

1. Individual. In the individual condition, participants will not be part of a team. They will receive weekly email feedback on their Walkstation performance (e.g. number of time slots they signed up for, and number of times they showed up for the time slot.) Participants will also receive a wellness tip in each email. (see appendix for a sample email)
2. Pairs. In the pair condition, participants will be randomly assigned to a partner. They will receive the same feedback as those in the individual condition, for both themselves AND their partner.
3. Group. In the group condition, participants will be randomly assigned to a group of 5 people. They will receive the same feedback as those in the individual condition, for both themselves AND each member of their group.

ELIGIBILITY:
Inclusion Criteria:

* Must pass the ParQ
* Must be employee of BCBS Massachusetts

Exclusion Criteria:

* Failing the ParQ
* Not being an employee of BCBS Massachusetts

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2010-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
WalkStation usage | 3 months
  Frequency with which the participant uses the WalkStation

SECONDARY OUTCOMES:
Creativity | 3 months
  Creativity measured on versus off the WalkStation.
Focus | 3 months
  Focus, as measured when person is on versus off the WalkStation.
Health Behaviors Survey | pre-baseline
  Survey of health-related behaviors to be completed by participant.
WalkStation Usage | 6 months
  Frequency with which the participant uses the WalkStation
Health Behaviors Survey | baseline
  Survey of health-related behaviors to be completed by participant.
Health Behaviors Survey | 6 months
  Survey of health-related behaviors to be completed by participant.
Creativity | baseline
  Creativity measured on versus off the WalkStation.
Focus | baseline
  Focus, as measured when person is on versus off the WalkStation.

CONTACTS AND LOCATIONS:
Locations (1):
- Blue Cross Blue Shield Massachusetts, Boston, Massachusetts, United States